CLINICAL TRIAL: NCT06685744
Title: Effectiveness of TeleNEUROrehabilitation Systems for Timely and Personalized Interventions and Vigilant Care in Neurodegenerative Conditions: the FIT4TeleNEURO Pragmatic Trial
Brief Title: TeleNEURO-Rehabilitation Systems for Neurodegenerative Conditions: the FIT4TeleNEURO Pragmatic Trial
Acronym: FIT4TeleNEURO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Collaborators: Fondazione Don Carlo Gnocchi Onlus, IRCCS Milano (Unknown); Fondazione Don Carlo Gnocchi Onlus, Centro S Maria della Provvidenza, Roma (Unknown); Fondazione Mondino (Other); Istituti Clinici Scientifici Maugeri SpA, IRCCS Bari (Unknown); Istituti Clinici Scientifici Maugeri SpA, IRCCS Pavia (Unknown); Istituti Clinici Scientifici Maugeri SpA, IRCCS Milano (Unknown); Istituti Clinici Scientifici Maugeri SpA, IRCCS Montescano (Unknown); Istituti Clinici Scientifici Maugeri SpA, IRCCS Telese (Unknown); IRCCS Azienda Ospedaliera Universitaria San Martino - Genova (Unknown); University of Modena and Reggio Emilia (Other); Centro Riabilitativo Villa Beretta (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FIT4TeleNEURO
Record Dates: First submitted 2024-10-29; First posted 2024-11-12 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2024-11

CONDITIONS: Parkinson Disease; Multiple Sclerosis; Neurologic Diseases, General
Keywords: Telerehabilitation; Digital Medicine; Chronic Neurological diseases; Rehabilitation; Telemedicine; Parkinson's Disease; Multiple Sclerosis; ehealth
MeSH Terms: conditions — Parkinson Disease; Multiple Sclerosis; Nervous System Diseases

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- TRsA (Experimental): Telerehabilitation (TR) single Approach - TRsA
  Interventions: Device: Telerehabilitation_TRsA
- TRcA (Experimental): Telerehabilitation (TR) combined Approach - TRcA
  Interventions: Device: Telerehabilitation_TRcA
- ET (Placebo Comparator): Educational treatment - ET
  Interventions: Behavioral: Educational treatment

INTERVENTIONS:
Device: Telerehabilitation_TRsA — Frequency: 5 weeks (4 sessions/week) of Telerehabilitation intervention provided according to a mixed model (3 asynchronous sessions + 1 synchronous session/week); Intensity: customized according to the patient's functional abilities (system's feedback); Time: 50 minutes/session; Type: exercises aimed at improving functional mobility and physical capacity according to a Task-oriented approach.
  Other Names: Telemedicine; Digital Medicine
  Arms: TRsA
Behavioral: Educational treatment — Home rehabilitation indications according to a conventional approach, customized according to the disease.
  Other Names: Placebo treatment
  Arms: ET
Device: Telerehabilitation_TRcA — Frequency: 5 weeks (4 sessions/week) of Telerehabilitation intervention provided according to a mixed model (3 asynchronous sessions + 1 synchronous session/week); Intensity: customized according to the patient's functional abilities (system's feedback); Time: 50 minutes/session; Type: a combination of exercises aimed at improving functional mobility and physical capacity according to a Task-oriented approach together with exercises aimed at recovering muscle strength (resistance) and improving endurance (endurance) using an Impairment-oriented approach.
  Other Names: Telemedicine; Digital medicine
  Arms: TRcA

SUMMARY:
The goal of the FIT4TeleNEURO pragmatic trial is to verify, in real-life care contexts, the superiority in terms of the effectiveness of early rehabilitation intervention with Telerehabilitation (TR) protocols (TR single Approach, task-oriented - TRsA; TR combined approach, task-oriented and impairment-oriented - TRcA) compared to conventional management (Educational treatment, ET).

The main questions it aims to answer are:

* Are Telerehabilitation protocols more effective than educational treatment?
* Is the TRcA treatment more effective than the TRsA? The study investigates the effects of rehabilitation treatment by comparing the two target cases (Multiple Sclerosis - MS and Parkinson's Diseases - PD).

Participants will be subjective to:

* 3 time-point of assessment (baseline, post-treatment and follow up) with motor, cognitive and quality-of-life measures
* A 5-weeks rehabilitation treatment (4 times/week)

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of probable PD according to MDS criteria (Postuma et al., 2015) in staging between 1 and 3 on the Hoehn & Yahr scale (Goetz et al., 2004) or diagnosis of MS according to the criteria of MC Donald 2010 (Polman et al., 2011) with disability level at the Expanded Disability Status Scale EDSS (Kurtzke, 1983) ≤ 4.5;
* age between 25 and 85 years;
* preserved cognitive level at the Montreal Cognitive Assessment test (MoCA test >15.5) (Santangelo et al., 2015);
* no rehabilitation program in place at the time of enrolment;
* stable drug treatment (last three month) with L-Dopa or dopamine agonists (PD group) or Disease Modifying Therapies (DMTs) (MS group).

Exclusion Criteria:

* presence of comorbidities that might prevent patients from undertaking a safe home program or determining clinical instability (i.e., severe orthopedic or severe cognitive deficits);
* presence of major psychiatric complications or personality disorders;
* presence of severe impairment of visual and/or acoustic perception;
* falls resulting in injuries or more than 2 falls in the 6 months prior to recruitment (PD and MS groups).
* pregnancy
* relapse ongoing/at least 3 months since the last relapse (MS group);
* presence of "frequent" freezing as recorded at the administration of Section II (daily life activity) of the UPDRS (score ≥ 3) (PD group);
* EDSS-FS (cerebellar function) ≥ 3 (MS group).

Ages: 25 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Change in static and dynamic balance as measured by the Mini-Best Test | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The Mini-BESTest aims to identify the disordered systems underlying the postural control responsible for poor functional balance. This tool is composed by 27 tasks (36 items in total) assessing bio-mechanical constraints, stability limits/verticality, anticipatory responses, postural responses, sensory orientation, and stability in gait. Each item is scored based on ordinal scale scoring from 0- 3 where 3 = best performances and 0 = worst performances. The total score is provided as a percentage. Higher scores are indicative of better performance.

SECONDARY OUTCOMES:
Change in dynamic and static balance measured by the Fullerton Advanced Balance Scale - FAB | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The FAB Scale evaluates dynamic and static balance under different situations. The test consists of 10 items that assess different aspects of balance, such as standing with eyes closed, reaching forward, turning, stepping, and standing on one leg. Each activity is scored on a 5-point scale from 0 to 4, where higher scores indicate better performance. The total score ranges from 0 to 40, with a score of 25 or lower indicating balance disturbances.
Change in dynamic balance as measured by the modified Dynamic Gait Index - mDGI | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The mDGI measures the capacity to adapt gait to complex tasks utilizing 8 tasks and 3 facets of performance (gait pattern score [0 -3], level of assistance [0 -2], and time level score [0 -3]). The total task score (range 0 -8) is calculated by summing the 3 performance facet scores for each task. Higher scores are indicative of better performance.
Change in perceived stability during activities of daily living as measured by the Activities Balance Confidence scale - ABC | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  ABC is a 16-item questionnaire that measures an individual's confidence during activities without falling or experiencing a sense of unsteadiness. Each item is scored ranging from 0 to 100. Higher scores are indicative of higher perceived stability.
Change in perceived fatigue during activities of daily living measured by the Fatigue Severity Scale - FSS | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The FSS questionnaire contains nine items that rate the severity of your fatigue symptoms on daily-life activities. Each item is scored ranging from 1 to 7. Higher scores are indicative of higher perceived fatigue.
Change in functional lower limbs strength as measured by the Five Times Sit to Stand Test - 5xSTS | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The 5xSTS asses functional lower limbs strength, transitional movements, balance, and fall risk. The scoring is based on the amount of time a patient is able to transfer from a seated to a standing position and back to sitting five times. The lower the time to complete the test, the better the outcome of the test.
Change in mobility and leg function performance as measured by the Timed 25 Foot Walk - T25FW | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The T25FW is a quantitative mobility and leg function performance test based on a timed 25 foot walk. The patient is directed to one end of a clearly marked 25 foot course and is instructed to walk 25 feet as quickly as possible. The time is calculated from the initiation of the instruction and ends when the patient has reached the 25 foot mark. The task is immediately administered again by having the patient walk back the same distance. The score is the average of the two completed trials.
Change in aerobic capacity and endurance as measured by the 6-Minute Walk Test - 6MWT | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The 6MWT assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity. An increase in the distance walked indicates improvement in basic mobility
Change in global cognitive functioning as measured by the Montreal Cognitive Assessment test - MoCA | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The MoCA test is a screening battery which also includes subtests to assess frontal functions such as set-shifting, abstraction and cognitive flexibility (MoCA total score range: 0-30). High scores are indicative of better general cognitive performance.
Change in visuoperceptual and attentional abilities as measured by the Trail Making Test - TMT parti A e B | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The TMT is a neuropsychological test that involves visual scanning (TMT-A) and dual-task (TMT-B). The TMT is scored by how long it takes to complete each part of the test. High execution times indicate poor performance.
Change in visuoperceptual and attentional abilities as measured by the Symbol Digit Modalities Test - SDMT, Smith A., 1973; Nocentini U., 2006 | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The SDMT is a commonly used test to assess psychomotor speed. This paper-pencil measure involves a substitution task using a coding key with nine different abstract symbols, each paired with a numeral. Below the key, a series of these symbols is presented, and the participant is asked to write down the corresponding number for each symbol. The score consists of the number of correct substitutions within 90 seconds. Higher scores indicate better performance.
Change in the perceived level of disability as measured by the World Health Organization disability assessment schedule 2.0 - WHODAS 2.0 | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  WHODAS 2.0 assesses the functioning and disability level in six domains (cognition, mobility, self-care, getting along, life activities, and participation in community activities) according to the International Classification of Functioning, Disability and Health (ICF). The summary scores for the WHODAS 2.0 will be obtained through 3 steps: 1) summing of item scores within each domain; 2) summing all six domain scores; 3) converting the summary score into a metric ranging from 0 to 100 (where 0 = no disability and 100 = full disability).
Change in depressive symptoms as measured by the Beck Depression Inventory - BDI-II | Baseline, 5 weeks after baseline, and follow-up (3 months after the end of treatment)
  The BDI-II is a 21-item questionnaire with each item rated on a 4-point scale (0-3). It is scored by summing ratings for each item (range 0-21). Higher scores indicate greater deflection of mood tone.

OTHER OUTCOMES:
System Usability Scale - SUS | 5 weeks after baseline
  The SUS is a 10 items questionnaire evaluating the perceived usability of a technological system or device. Each item is scored on a Likert scale from 0 to 5, and the total score range from 0 to 100. Higher scores are indicative of higher perceived usability.
Technology Acceptance Model - TAM3 | 5 weeks after baseline
  The TAM3 questionnaires evaluates the user acceptance of technology across 16 domains. Scoring is based on a Likert scale (from 1 = Strongly Disagree to 7 = Strongly Agree) or a 10-point Guttman scale. Higher scores are indicative of higher acceptance of technology.
Barthel Index | Baseline
  The Barthel Index is a scale used to measure a person's ability to perform basic activities of daily living (ADLs) independently. It evaluates 10 functions such as feeding, bathing, dressing, toileting, mobility, and stair climbing. Each activity is scored based on the level of assistance required, with a total score ranging from 0 (completely dependent) to 100 (completely independent).

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Istituti Clinici Scientifici Maugeri SpA, Bari
  - IRCCS Azienda Ospedaliera Universitaria San Martino, Genova
  - Centro Riabilitativo Villa Beretta, Lecco
  - Fondazione Don Carlo Gnocchi Onlus, IRCCS, Milan
  - University of Modena and Reggio Emilia, Modena
  - Istituto Neurologico Nazionale IRCCS Casimiro Mondino, Pavia

IPD SHARING:
Plan to Share IPD: Yes
all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: October 2024- December 2036
Access Criteria: Contact the principal investigator